CLINICAL TRIAL: NCT03847441
Title: Topical Calcipotriol Versus Narrowband Ultraviolet B in Treatment of Alopecia Areata: A Randomized Controlled Trial
Brief Title: Topical Calcipotriol Versus Narrowband Ultraviolet B in Treatment of Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Moustafa A. El Taieb, Head of Dermatology, Venereology and Andrology Department, Ass. Prof. Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Alopecia Calcipotiol
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Calcipotriol; Narrow Band-UVB; Vitamin D3
MeSH Terms: conditions — Alopecia Areata | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator)
  Interventions: Drug: Calcipotriol; Diagnostic Test: vitamin D3 level
- Group II (Active Comparator)
  Interventions: Device: Narrow Band UVB; Diagnostic Test: vitamin D3 level
- Group III (Active Comparator)
  Interventions: Drug: Calcipotriol; Device: Narrow Band UVB; Diagnostic Test: vitamin D3 level
- Group IV (Placebo Comparator)
  Interventions: Diagnostic Test: vitamin D3 level

INTERVENTIONS:
Drug: Calcipotriol — Calcipotriol ointment (0.005%)
  Arms: Group I; Group III
Device: Narrow Band UVB — NB-UVB (311nm) phototherapy
  Arms: Group II; Group III
Diagnostic Test: vitamin D3 level — vitamin D3 (ng/ml)

SUMMARY:
Alopecia Areata is a common condition. This study investigated the efficacy of calcipotriol versus Narrow Band Ultraviolet B in treatment of Alopecia areata and their effects on serum vitamin D3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Alopecia Areata of scalp

Exclusion Criteria:

Other causes of alopecias including scarring alopecia, androgenic alopecia, telogen effluvium autoimmune diseases, pregnant and lactating females

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of Alopecia Areata After treatment As assessed by Severity of Alopecia tool (SALT) score | 3 months
  calculation of SALT score before and after treatment
Improvement of serum Vitamin D levels in (ng/ml) after treatment | 3 months
  measurement of serum vitamin D before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No